CLINICAL TRIAL: NCT01010451
Title: Survival of Primary Molars Treated With Antimicrobial Pulpotomy or Calcium Hydroxide Pulpectomy
Brief Title: Antimicrobial Pulpotomy of Primary Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Universidade Federal de Goias, Dental School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3222
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Inflammation; Necrosis
Keywords: pulpotomy; pulpectomy; primary teeth; dental care for children
MeSH Terms: conditions — Inflammation; Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antimicrobial pulpotomy (Experimental): Pulpotomy of primary molars with pulp inflammation or necrosis due to carious lesions using an antimicrobial paste
  Interventions: Procedure: Antimicrobial pulpotomy
- Calcium hydroxide pulpectomy (Active Comparator): Pulpectomy of primary molars with pulp inflammation or necrosis due to carious lesions using a calcium hydroxide paste as intracanal medication
  Interventions: Procedure: Calcium hydroxide pulpectomy

INTERVENTIONS:
Procedure: Antimicrobial pulpotomy — Pulpotomy of inflamed or necrotic pulp using an antimicrobial paste (chloramphenicol, tetracycline, zinc oxide/eugenol)as medication.
  Other Names: Antibacterial pulp therapy; Antibacterial pulpotomy; Non-vital pulpotomy
  Arms: Antimicrobial pulpotomy
Procedure: Calcium hydroxide pulpectomy — Pulpectomy of inflamed or necrotic pulp using a calcium hydroxide paste as medication
  Arms: Calcium hydroxide pulpectomy

SUMMARY:
There is a lack of evidence of the long-term successful outcomes of antimicrobial endodontic treatment for primary teeth. This study intended to evaluate (by survival analysis) the effectiveness of an antimicrobial pulpotomy (chloramphenicol, tetracycline, zinc oxide/eugenol) in primary molars compared to calcium hydroxide pulpectomy, testing the hypothesis that antimicrobial pulpotomy could be an alternative pulp therapy for primary teeth with pulp inflammation or necrosis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children (ASA PS 1)
* Children presenting one or more primary molar with pulp inflammation or necrosis due to carious lesion and indicated for endodontic therapy

Exclusion Criteria:

* Lost to follow-up

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-08; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dental School, Goiânia, Goiás, Brazil